CLINICAL TRIAL: NCT02494024
Title: A Double-Blind, Placebo Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of C2N-8E12 in Subjects With Progressive Supranuclear Palsy
Brief Title: Safety, Tolerability, and Pharmacokinetics of C2N-8E12 in Subjects With Progressive Supranuclear Palsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C2N Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C2N-8E12-WW-104
Record Dates: First submitted 2015-06-30; First posted 2015-07-10 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Progressive Supranuclear Palsy
Keywords: PSP; C2N-8E12; tauopathy; Progressive Supranuclear Palsy; Steele Richardson Olszewski Syndrome; Humanized anti-tau antibody
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Tauopathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Single dose C2N-8E12 level 1 (Experimental): Single IV infusion of C2N-8E12
  Interventions: Drug: Single dose C2N-8E12
- Single dose C2N-8E12 level 2 (Experimental): Single IV infusion of C2N-8E12
  Interventions: Drug: Single dose C2N-8E12
- Single dose C2N-8E12 level 3 (Experimental): Single IV infusion of C2N-8E12
  Interventions: Drug: Single dose C2N-8E12
- Single dose C2N-8E12 level 4 (Experimental): Single IV infusion of C2N-8E12
  Interventions: Drug: Single dose C2N-8E12
- Single dose placebo (Placebo Comparator): Single IV infusion of placebo
  Interventions: Drug: Single dose placebo

INTERVENTIONS:
Drug: Single dose C2N-8E12 — C2N-8E12 is a humanized recombinant anti-human tau antibody.
  Arms: Single dose C2N-8E12 level 1; Single dose C2N-8E12 level 2; Single dose C2N-8E12 level 3; Single dose C2N-8E12 level 4
Drug: Single dose placebo — Subjects will be block randomized to receive a single dose of C2N-8E12 or placebo in two blocks of 4 subjects (3:1, C2N-8E12:placebo) per cohort.
  Arms: Single dose placebo

SUMMARY:
This study will evaluate the safety and tolerability (maximum tolerated dose (MTD) within the specified dosing range) of single intravenous (IV) infusion of C2N-8E12 in patients with progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
This study evaluates the safety, tolerability, pharmacokinetics, and maximum tolerated dose (within dosing range) of intravenous (IV) infusion of C2N-8E12 in 32 patients with progressive supranuclear palsy (PSP). Four sequential cohorts will receive increasing single doses of either C2N-8E12 or placebo. Out of every 4 patients enrolled 3 patients will receive drug and 1 will receive placebo. Study participants will be followed for a minimum of 2 months post-treatment to monitor for the safety, tolerability, pharmacokinetics, and immunogenicity of C2N-8E12.

ELIGIBILITY:
Key Inclusion Criteria:

* Meets NINDS-SPSP possible or probable criteria as modified for NNIPPS and AL-108-231 clinical trials
* Brain MRI at Screening is consistent with PSP;
* Stable medications for Parkinsonism for at least 2 months prior to Screening;
* Agree to use protocol specified methods of contraception.

Key Exclusion Criteria:

* Signs of a progressive neurological disorder that better meets the criteria for types of neurological disorders other than PSP;
* Currently on any other biologic or immunomodulatory therapy;
* Subjects that reside at a skilled nursing or dementia care facility;
* Diagnosis of any other significant unrelated neurological or psychiatric disorders that could account for cognitive deficits;
* Untreated major depression at baseline evaluation, based on clinical judgment and results in geriatric depression scale;
* Unable to tolerate MRI scan at Screening or any other contraindication to MRI;
* Any contraindication to or unable to tolerate lumbar puncture at Screening, including use of anti-coagulant medications.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by number of participants experiencing adverse events (AEs), serious AEs, and abnormalities in clinical laboratory tests, vital signs, ECGs, MRI, and physical and neurological exams. | up to 4 months

SECONDARY OUTCOMES:
Immunogenicity as measured by the number of participants developing anti drug antibodies. | up to 4 months
Area under the concentration vs time curve (AUC) of C2N-8E12 | up to 4 months
Elimination half-life of C2N-8E12 | up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — UCSF Memory and Aging Center
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - UCSD Department of Neurosciences, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Health Presbyterian Dallas, Dallas, Texas

REFERENCES:
- [Background] Yanamandra K, Kfoury N, Jiang H, Mahan TE, Ma S, Maloney SE, Wozniak DF, Diamond MI, Holtzman DM. Anti-tau antibodies that block tau aggregate seeding in vitro markedly decrease pathology and improve cognition in vivo. Neuron. 2013 Oct 16;80(2):402-414. doi: 10.1016/j.neuron.2013.07.046. Epub 2013 Sep 26. PMID 24075978
- [Background] Boxer AL, Lang AE, Grossman M, Knopman DS, Miller BL, Schneider LS, Doody RS, Lees A, Golbe LI, Williams DR, Corvol JC, Ludolph A, Burn D, Lorenzl S, Litvan I, Roberson ED, Hoglinger GU, Koestler M, Jack CR Jr, Van Deerlin V, Randolph C, Lobach IV, Heuer HW, Gozes I, Parker L, Whitaker S, Hirman J, Stewart AJ, Gold M, Morimoto BH; AL-108-231 Investigators. Davunetide in patients with progressive supranuclear palsy: a randomised, double-blind, placebo-controlled phase 2/3 trial. Lancet Neurol. 2014 Jul;13(7):676-85. doi: 10.1016/S1474-4422(14)70088-2. Epub 2014 May 27. PMID 24873720
- [Background] Litvan I, Agid Y, Calne D, Campbell G, Dubois B, Duvoisin RC, Goetz CG, Golbe LI, Grafman J, Growdon JH, Hallett M, Jankovic J, Quinn NP, Tolosa E, Zee DS. Clinical research criteria for the diagnosis of progressive supranuclear palsy (Steele-Richardson-Olszewski syndrome): report of the NINDS-SPSP international workshop. Neurology. 1996 Jul;47(1):1-9. doi: 10.1212/wnl.47.1.1. PMID 8710059
- [Background] Yanamandra K, Jiang H, Mahan TE, Maloney SE, Wozniak DF, Diamond MI, Holtzman DM. Anti-tau antibody reduces insoluble tau and decreases brain atrophy. Ann Clin Transl Neurol. 2015 Mar;2(3):278-88. doi: 10.1002/acn3.176. Epub 2015 Jan 23. PMID 25815354